CLINICAL TRIAL: NCT06658067
Title: CGMs for All: Studying the Impact of Expanding CGM Access
Brief Title: Continuous Glucose Monitors (CGMs) for All: Studying the Impact of Expanding CGM Access
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Yale Office of Global Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000038335
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Type 2 Diabetes; Type 2 Diabetes Mellitus - Poor Control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Poorly Controlled Type 2 Diabetes- CGM (Experimental): Participants will have CGM sensor placed at first visit and will be worn for 12 weeks. Sensor must be scanned 3 times daily. Adjustments to medication regimen will be recommended at 6 weeks. Follow-up appointments will be at 12 weeks and 24 weeks.
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — The first CGM sensor will be applied as directed during the first visit with a brief training by staff. Participant will be instructed to remove and replace the device every 14 days for the remainder of the 3-month trial period. Participant will also be instructed to scan the sensor three times daily. Compliance may be tracked via remote accessing of the blood glucose log on the online FreeStyle portal. CGM models used will include the Abbott FreeStyle Libre 2 and 3 and Dexcom G5, G6 and G7.

SUMMARY:
This non-blinded, non-randomized pre-post study will examine the impact of providing CGM sensors free of charge to adult patients of Fair Haven Community Health Care with poorly controlled type 2 diabetes on glycemic control and quality of life.

DETAILED DESCRIPTION:
This study will enroll adult patients with type 2 diabetes and A1c of 8.0 or greater despite long-term use of insulin who are underinsured and under-resourced , meaning they are unable to reasonably afford CGM sensors. The participants will be chosen from among the panels of three providers.

This study aims to determine whether providing CGMs free of charge to patients with poorly controlled diabetes who could not otherwise afford them positively impacts their glycemic control and quality of life.

FHCHC's clinicians will identify adult patients from their panel with type 2 diabetes and poor glycemic control (A1c at least 8) on insulin who may be unable to afford CGM. Once consented, participants will have point-of-care A1c testing as well as pregnancy testing (if applicable); patient eligibility based on glycemic control criterion should be determined by this A1c. Participants will then complete the study questionnaires. Clinic staff will teach CGM sensor placement and determine whether a reader is required or if a compatible mobile device for intermittent scanning will be used. Blood Glucose (BG) readings are provided via online Libre portal.

At the 6-week follow-up visit, the provider will recommend adjustments to the participant's medication regimen based on their BG trends on CGM and their clinical judgment. Providers will ask participants to report any adverse events, safety issues, or trouble with the CGM system thus far experienced.

At the 12-week follow-up visit, participants will repeat completion of study questionnaires and undergo second A1c measurement. Further adjustment to medication regimen is permitted as provider sees fit.

At the 24-week follow-up visit, participants will repeat completion of study questionnaires for a third time and undergo third A1c measurement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with type 2 diabetes mellitus
* A1c greater than or equal to 8.0 within two weeks of the time of enrollment
* On insulin for at least one year +/- other antihyperglycemics
* Ability and willingness to wear CGM for 14-day periods throughout the trial period
* Ability and willingness to comply with provider-directed adjustments to medication regimen
* Inability to afford CGM sensors

A note on Vulnerable Populations: Many of FHCHC's patients are economically disadvantaged and of minority backgrounds; the clinic's patient base may be considered to constitute a vulnerable population. As such, recruitment and enrollment will be conducted within a vulnerable population. The nature of the study requires this, and the results are intended to directly benefit this population through the potential for improved glycemic control and quality of life.

Exclusion Criteria:

* Insulin naïve
* Diabetic ketoacidosis (DKA) in previous 6 months
* End-Stage Renal Disease (ESRD)
* Contraindications to CGM use
* Active insurance plan that would provide enough of a subsidy for participant to feasibly purchase CGM sensors
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean Illness Intrusiveness Ratings Scale score (IIRS) | Baseline, 12 weeks, 24 weeks
  The IIRS is a useful, easy-to-apply tool that measures the degree of illness-induced disruptions in the 13 different aspects of life. Total score range from 13 (minimal intrusiveness) to 91 (extreme intrusiveness).
Mean Hemoglobin A1c concentration | Baseline, 12 weeks, 24 weeks
  Mean A1c concentration in mg/dL measured in blood samples

SECONDARY OUTCOMES:
Mean Treatment Burden Questionnaire (TBQ) score | Baseline, 12 weeks, 24 weeks
  The TBQ is composed of 13 items rated on a Likert scale ranging from 0 (not a problem), to 10 (big problem). Item scores can be summed into a total score, ranging from 0 to 130. Higher scores indicate higher burden.
Mean Diabetes Distress Scale score (DDS-17) | Baseline, 12 weeks, 24 weeks
  DDS-17 is a 17-item measure that uses a Likert scale with each item scored from 1 (no distress) to 6 (serious distress) concerning distress experienced over the last month. Total score range from 1 to 6 with higher scores indicating more distress.
Mean Summary of Diabetes Self-Care Activities (SDSCA) score | Baseline, 12 weeks, 24 weeks
  The SDSCA is a brief self-report questionnaire of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking.Total score range is 7-70. Higher scores indicate more days spent doing diabetes self-care activities (such as checking blood sugar, following a diet plan, and participating in exercise activities).
Score on digital supplement to TBQ (TBQ+D) | Baseline, 12 weeks, 24 weeks
  The TBQ+D adds an additional 6 items to the TBQ, each rated on a Likert scale ranging from 0 (not a problem) to 10 (big problem). Item scores can be summed into a total score, ranging from 0 to 60. Higher scores indicate higher burden incurred by the use of digital health devices.
Quality of life analogue scale | Baseline, 12 weeks, 24 weeks
  This scale asks respondents to rate how diabetes has affected their quality of life over the last 2 weeks on a scale from 0 (the worst it has ever been) to 10 (the best it has ever been). Higher scores indicate better perceived quality of life.
TBQ+D Cognitive Interview tool | Baseline, 12 weeks, 24 weeks
  Cognitive Interview Tool: 10 participants will be asked to complete the TBQ+D survey aloud and provide their thoughts about the questions included. These recordings will be transcribed and evaluated qualitatively for recurrent themes.

CONTACTS AND LOCATIONS:
Overall Officials: Kasia Lipska, MD MHS, Principal Investigator — Yale University
Locations (1):
- Fair Haven Community Health Care (FHCHC), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual study data for the participants completing the Cognitive Interview Tool will be deidentified and shared with collaborators at the Mayo Clinic. Investigators have completed a Data Usage Agreement (DUA) with the Yale Office of Sponsored Projects (OSP).